CLINICAL TRIAL: NCT05409547
Title: A Multi-center, Open, Randomized, Controlled Clinical Study of Autologous Peripheral Blood Stem Cell Mobilization for Pegylated Recombinant Human Granulocyte Colony Stimulating Factor
Brief Title: A Clinical Study of Autologous Peripheral Blood Stem Cell Mobilization for PEG-G-CSF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ning Huang (Other)
Responsible Party: Sponsor-Investigator, Ning Huang, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YKLL-KY-2022(009)
Record Dates: First submitted 2022-05-24; First posted 2022-06-08 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Granulocyte Colony-stimulating Factor; Stem Cell Mobilization
Keywords: Hematopoietic stem cell mobilization; Hematopoietic stem cell transplantation; pegylated granulocyte colony-stimulating factor
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-G-CSF (Experimental): 6 mg, single dose
  Interventions: Drug: PEG-rhG-CSF
- rhG-CSF (Active Comparator): 5 μg/kg, twice a day
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — PEG-rhG-CSF 6 mg/d (single dose) will be given on the second day after chemotherapy.
  Other Names: rhG-CSF

SUMMARY:
Have a comparison between pegylated recombinant human granulocyte colony stimulating factor (PEG-rhG-CSF) and recombinant human granulocyte-colony stimulating factor (rhG-CSF) for difference in efficacy of hematopoietic reconstruction after autologous peripheral blood stem cell mobilization (PBSCM) and autologous peripheral blood stem cell transplantation (APBSCT).

Primary purpose:

Compare the difference between PEG-rhG-CSF and G-CSF in PBSCM.

Secondary purpose:

Compare the difference between PEG-rhG-CSF and G-CSF in APBSCT.

DETAILED DESCRIPTION:
Key issues to be addressed:

To compare the efficiency of stem cell mobilization and hematopoietic system reconstruction between PEG-rhG-CSF and rrhG-CSF.

Research design:

A multicenter, open, prospective randomized controlled clinical study.

Research objects:

Patients with hematological diseases who will receive autologous hematopoietic stem cell mobilization (including lymphoma, myeloma patients who achieved PRand MRD-negative acute leukemia patients ).

Number of cases:

There will be 40 cases in the treatment group and the control group, respectively. The cases will be randomly divided into PEG-rhG-CSF or rhG-CSF control group to receive treatment. The cases will be assigned to 1 experimental group and 1 control group in a 1:1 ratio.

Experiment design Overall design A multicenter, randomized, open-controlled study will be used. We will include patients who meet the indications of autologous hematopoietic stem cell transplantation as the research objects. Chemotherapy will be given prior to mobilization: chemotherapy regimens will be given to patients before mobilization according to the type of disease (such as etoposide alone, cyclophosphamide alone, VP-16+ CTX, medium-dose cytarabine, etc.). The experimental group will receive subcutaneous injection of PEG-rhG-CSF (6 mg) once on the 2nd day after chemotherapy. For the control group, the peripheral blood changes will be closely monitored after chemotherapy, and rhG-CSF (5 μg/kg/d) will be applied twice a day at the beginning of the leukocyte rising phase until the acquisition ends. The patients who meet the requirements for enrollment will be randomly divided into the experimental group and the control group in a 1:1 ratio.

Total number of cases This phase of the clinical trial will include patients who meet the indications for autologous hematopoietic stem cell transplantation as the research subjects, and the included patients will be randomly divided into different-dose PEG-rhG-CSF group or rhG-CSF control group to receive treatment. This trial plans to enroll 80 patients and assign them to 1 experimental group and 1 control group in a 1:1 ratio.

Dose for mobilization

Experimental group:

PEG-rhG-CSF 6 mg/d (single dose) will be given on the second day after chemotherapy. Routine peripheral blood test and CD34+ cell count will be done 1 day before collection.

Control group:

rhG-CSF (5 μg/kg/d) will be given twice a day, and peripheral blood stem cells will be collected on the 5th day. Routine peripheral blood test and CD34+ cell count will be done 1 day before collection. rhG-CSF (5 μg/kg/d) twice a day could be temporarily added if CD34+ cell count is less than 20/μL.

Collection of stem cells:

Stem cells will be collected by a blood cell separator. If the number of CD34+ collected on the first day is not enough, the collection will continue on the second day, with a collection time ≤5 hours. Judgment of collection results: ①Successful collection: the number of CD34+ cells obtained in one collection is ≥2×10^6/kg; ②Failure of collection: the number of CD34+ cells obtained by 3 collections is less than 2×10^6/kg; ③ Excellent collection: the number of CD34+ cells obtained in one collection is ≥5×10^6/kg.

Preconditioning scheme All transplant patients will receive preconditioning therapy according to their disease type.

Stem cell reinfusion Hematopoietic stem cells will be reinfused for all cases 24 hours after the end of preconditioning therapy. The total amount of hematopoietic stem cells reinfused in each group: MNC≥4.0×10^8/kg, and CD34+ cells≥2.0×10^6/kg. The actual volume of reinfusion of each group will be recorded.

Hematopoietic reconstitution criteria After reinfusion of hematopoietic stem cells, if blood cells continue to decline and then rise again, and neutrophils exceed 0.5×10^9/L for 3 consecutive days, the leukocyte reconstitution criteria are met; In the absence of platelet transfusion, if platelet count is greater than 20×10^9/L for 3 consecutive times, the platelet reconstitution criteria are met.

Experimental drug:

PEG-rhG-CSF vs. rhG-CSF.

Promotion of bone marrow reconstruction:

Starting on the 4th day after hematopoietic stem cell reinfusion, rhG-CSF will be administered at a dose of 5μg/kg/d until the granulocytes rise to more than 5000/ul and become stable.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as hematological diseases definitely, body weight ≥30kg, age: 18-60 years, without limitation in gender or race;
2. Patients who receive APBSCT voluntarily;
3. Patients who participate in the open randomized controlled study of autologous hematopoietic stem cell mobilization for PEG-rhG-CSF and G-CSF voluntarily;
4. Each subject must sign the informed consent from (ICF) to indicate that he/she understands the purposes and procedures of the study, and participates in the study voluntarily. Considering the patient's conditions, if the patient's signature is not conducive to treatment, his/her legal representative will sign the ICF.

Exclusion Criteria:

1. Patients who have serious organ dysfunctions or diseases, such as serious diseases or dysfunctions heart, liver, kidney, pancreas and etc.;
2. Patients who cannot tolerate autologous hematopoietic stem cell transplantation and autologous stem cell mobilization;
3. Subjects who and/or whose authorized family members refuse HSCT or PEG-rhG-CSF treatment;
4. Subjects with any life-threatening disease, medical condition or organ system dysfunction compromising their safety or causing unnecessary risks for the study results in the investigator' opinion, with drug dependence, with uncontrolled mental illness, or with cognitive dysfunction;
5. Subjects who participate in other similar clinical studies within 3 months;
6. Subjects who are considered as unsuitable for the study by the investigator (e.g., those expected to be unable to adhere to relevant treatment regimen due to financial problems).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Efficiency of stem cell mobilization | 3years
  Count of collected CD34+ cells (CD34+ > 2×10^6 /kg will be considered as successful mobilization).

SECONDARY OUTCOMES:
Time of hematopoietic reconstitution | 3years
  1. The time period(days) between reinfusion of hematopoietic stem cells and neutrophils exceed 0.5×10^9/L for 3 consecutive days.
  2. The time period(days) between reinfusion of hematopoietic stem cells and platelet count is greater than 20×10^9/L for 3 consecutive times.

CONTACTS AND LOCATIONS:
Overall Officials: ning huang, Professor, Principal Investigator — professor; kehong bi, Professor, Study Director — professor